CLINICAL TRIAL: NCT00005563
Title: Multicenter Asthma Research Collaboration
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5110; R03HL063253 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2002-09

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To study the epidemiology of emergency asthma by focusing on three Multicenter Asthma Research Collaboration (MARC) databases collected over a two-year period in adult and pediatric emergency departments.

DETAILED DESCRIPTION:
BACKGROUND:

The Multicenter Airway Research Collaboration (MARC) was created by 12 emergency physicians in May 1996 to determine the best management of acute asthma in the emergency department. The principal investigator of MARC, Dr. Carlos Camargo, formed the MARC Steering Committee to help guide this collaboration. The MARC Coordinating Center is based at the Massachusetts General Hospital (Boston, MA). Financial support for MARC has come from a variety of sources, including government, foundations, and industry. The NHLBI study used MARC databases.

DESIGN NARRATIVE:

Five representative aims were to: 1) characterize acute asthma management in urban emergency departments (EDs) and then compare current practice with that recommended in the 1997 national guidelines; 2) examine gender differences in acute asthma; 3) identify reasons why minority patients with asthma go to (and possibly prefer) the ED for their asthma care; 4) characterize important clinical subgroups, such as acute asthma among pregnant women and patients with sudden-onset severe acute asthma; and 5) examine risk factors for asthma hospitalization and for relapse after ED discharge.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07; Study Completion 2001-06 (Actual)

REFERENCES:
- [Background] Emerman CL, Cydulka RK, Crain EF, Rowe BH, Radeos MS, Camargo CA Jr; MARC Investigators. Prospective multicenter study of relapse after treatment for acute asthma among children presenting to the emergency department. J Pediatr. 2001 Mar;138(3):318-24. doi: 10.1067/mpd.2001.111320. PMID 11241036
- [Background] Emond SD, Reed CR, Graff LG IV, Clark S, Camargo CA Jr. Asthma education in the Emergency Department. On behalf of the MARC Investigators. Ann Emerg Med. 2000 Sep;36(3):204-11. doi: 10.1067/mem.2000.109168. PMID 10969221